CLINICAL TRIAL: NCT06689540
Title: First-in-human Clinical Study of Mts105 for Advanced Hepatocellular Carcinoma
Brief Title: Mts105 for Advanced Hepatocellular Carcinoma
Acronym: MTS105 for HCC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shen Lin (Other)
Collaborators: METiS Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Shen Lin, Professor, Peking University
Organization: Peking University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MTS105-01
Record Dates: First submitted 2024-11-08; First posted 2024-11-14 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-10

CONDITIONS: Liver Cancer, Adult; Metastatic Liver Cancers; HCC - Hepatocellular Carcinoma; Hepatocellular Carcinoma (HCC)
Keywords: hcc; mts105; metis; mRNA; LNP
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: Bayesian Optimal Interval (BOIN) Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- dose level #1 (Experimental): Starting dose, 0.05 ug/kg
  Interventions: Biological: MTS105
- dose level #2 (Experimental): dose escalation, 0.5 ug/kg
  Interventions: Biological: MTS105
- dose level #3 (Experimental): dose escalation, 3.0 ug/kg
  Interventions: Biological: MTS105
- dose level #4 (Experimental): dose escalation, 15.0 ug/kg
  Interventions: Biological: MTS105
- dose level #5 (Experimental): dose escalation, 30.0 ug/kg
  Interventions: Biological: MTS105
- dose level #6 (Experimental): dose escalation, 45.0 ug/kg
  Interventions: Biological: MTS105

INTERVENTIONS:
Biological: MTS105 — MTS105 is a combination of mRNA, which encodes a therapeutic protein, and its delivery vehicle, a lipid nanoparticle (LNP). The starting dose is estimated based on the Minimal Anticipated Biological Effect Level (MABEL) derived from non-clinical studies.
  A starting dose of 0.05 μg/kg was proposed for this study; following dose strength for escalation are: 0.5 μg/kg, 3.0 μg/kg, 15 μg/kg, 30 μg/kg, 45 μg/kg.

SUMMARY:
This is the first-in-human trial of MTS105 (mRNA-LNP). The goal of this clinical trial is to evaluate the safety, tolerability of intravenous injection of MTS105 in advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
MTS105 is an mRNA-LNP combination. Once the mRNA is delivered to the liver via lipid nanoparticles (LNP), it translates into a therapeutic bispecific T-cell engager designed to activate T cells to target and destroy liver cancer cells.

MTS105 is anticipated to offer liver-targeted delivery, specific binding to hepatocellular carcinoma cells, a broad therapeutic window, and potent anti-tumor effects.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of hepatocellular carcinoma (HCC), excluding fibrolamellar or sarcomatoid subtypes, as well as mixed hepato-cholangiocellular carcinoma;
2. Positive for GPC3 expression per immunohistochemical (IHC) staining.
3. Failure of standard systemic therapies, including at least one immune checkpoint inhibitor and one targeted therapy (Tyrosine Kinase Inhibitors, and/or anti vascular endothelial growth factor agent).
4. Presence of a measurable tumor lesion (per RECIST/ mRECIST criteria).
5. Barcelona Clinical Liver Cancer Stage B or C (BCLC B/C)
6. Child-Pugh Score ≤ 6
7. ECOG score ≤ 1
8. Adequate organ and bone marrow function as defined by the following laboratory criteria:

   1. Hematology: No blood transfusion or colony-stimulating factor therapy within 7 days prior to the first dose. The following hematological parameters should be met:Absolute neutrophil count ≥ 1.5 × 10^9/L;Lymphocyte count ≥ 0.5 × 10^9/L;Hemoglobin ≥ 90 g/L;Platelet count ≥ 75 × 10^9/L;
   2. Liver function:Total bilirubin ≤ 2.5 mg/dL;Albumin ≥ 28 g/L;Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 × ULN;
   3. International Normalized Ratio (INR) ≤ 2.3;Oral anticoagulant therapy at a stable dose for at least 2 weeks. If oral warfarin is used, the patient must have an INR ≤ 3.0 and no bleeding events within 28 days prior to administration;
   4. Renal function:Serum creatinine ≤ 1.5 × ULN, or endogenous creatinine clearance ≥ 45 mL/min (as determined by the CKD-EPI formula);Urinary protein < 2+, or urinary protein ≥ 2+ but with 24-hour protein quantification ≤ 1.0 g
   5. Cardiac function:Left ventricular ejection fraction (LVEF) ≥ 50%; No clinically significant abnormal ECG findings (chronic atrial fibrillation is allowed, provided it does not require medication);
9. Capable of full communication with the investigator, with the ability to understand and comply with study requirements, and able to understand and sign the informed consent form (ICF).
10. ≥18 years

Exclusion Criteria:

1. Any known active intracranial metastases, or brain metastases that have been treated for less than 4 weeks.
2. Recent Antitumor Therapy:

   1. Treatment with any immune checkpoint inhibitor within 4 weeks (28 days) prior to the first dose.
   2. Received any investigational drug within 4 weeks prior to the first dose.
   3. Received localized therapy for hepatocellular carcinoma (HCC), including but not limited to arterial chemoembolization (TACE), arterial infusion chemotherapy (HAIC), Y-90 radioembolization, ablative therapy, or stereotactic radiation therapy (SBRT), within 4 weeks prior to the first dose.
   4. Received other anticancer therapies, such as multi-targeted tyrosine kinase inhibitors (mTKIs) and/or anti-VEGF therapies, within 3 weeks.
   5. Received non-specific immunomodulatory therapy, including but not limited to interleukin, interferon, thymidine, etc., within 2 weeks prior to the first dose.
   6. Received herbal or proprietary Chinese medicine for antitumor indications within 1 week prior to the first dose.
   7. Previously received experimental treatment targeting GPC3 (patients may be enrolled if they remain positive for GPC3 upon testing).
3. History of liver transplantation or hematopoietic stem cell transplantation.
4. Unresolved toxicity from prior anticancer therapy (> grade 1, according to CTCAE v5.0).
5. Major surgery (other than biopsy) within 28 days prior to the first dose.
6. Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 90 mmHg).
7. Class III-IV heart failure by New York Heart Association (NYHA) criteria within 6 months prior to the first dose, unstable angina, myocardial infarction, bypass surgery, stent placement, cerebral infarction, or clinically significant valvular heart disease.
8. QTcF ≥ 450 ms in men and ≥ 470 ms in women (by Fridericia formula).
9. Severe infection within 4 weeks before the first dose (excluding viral hepatitis), or any signs or symptoms of active infection within 2 weeks before the first dose, or patients requiring antibiotic treatment within 2 weeks (excluding local medications and prophylactic antibiotics); unexplained fever > 38.5°C before the first dose.
10. For HBV-associated HCC:

    1. HBsAg (+) : less than 2 weeks of HBV antiviral standard treatment before the first administration of study drug, with an HBV DNA viral load ≥ 1000 IU/mL.
    2. HBcAb (+) , HBsAg (-): HBV DNA viral load ≥ 1000 IU/mL.
11. Hepatitis C virus-infected subjects who have not completed 4 weeks of antiviral treatment.
12. Positive for human immunodeficiency virus (HIV+).
13. Subjects requiring systemic corticosteroids (equivalent dose of prednisone > 10 mg/day) or other immunosuppressive drugs within 14 days prior to the first dose or during the study.
14. History of autoimmune disease requiring systemic treatment within 2 years prior to the first dose.
15. History of other malignancies within 2 years prior to the first dose (excluding cured skin basal cell carcinoma or squamous cell carcinoma, cervical carcinoma in situ, breast ductal carcinoma in situ, or other cancers that the investigator believes are cured and have an extremely low risk of recurrence).
16. Women who are pregnant or breastfeeding.
17. Any other condition that, in the opinion of the investigator, makes participation in the study inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), and serious adverse events (SAEs). | From enrollment to the end of treatment at 4 weeks
  Incidence of TEAEs,and SAEs.
Maximal Tolerance Dose (MTD) | Within the first 28-days following first dose
  Determined based on the occurrence of dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Within the first 28-days following first dose
  Peak Plasma Concentration of the investigational product
Area under the plasma concentration versus time curve (AUC) | Within the first 28-days following first dose
Time for peak concentration (Tmax) | Within the first 28-days following first dose
  Time for peak concentration
Elimination half-life | Within the first 28-days following first dose
  Elimination rate of the therapeutic protein in circulation.
Steady-state concentration | Within the first 28-days following first dose
  steady-state concentration
Objective Response Rate | through study completion, an average of 1 year
  The proportion of participants who have a confirmed CR or confirmed PR as determined by the investigator at local site per RECIST v1.1 or mRECIST 1.1
Duration of Response (DOR) | through study completion, an average of 1 year
  The time from first documented confirmed response until date of documented progression of disease, as determined by investigator at local site or death due to any cause.
Progression Free Survival (PFS) | through study completion, an average of 1 year
  Time from infusion date until progression, as assessed by the investigator at local site, or death due to any cause.
Overall Survival (OS) | through study completion, an average of 1 year
  Overall Survival (OS)

OTHER OUTCOMES:
Concentration of anti-drug antibodies | through study completion, an average of 1 year
  Immunogenicity, anti-drug antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No